CLINICAL TRIAL: NCT05195827
Title: Evaluation of Once-Daily PRM125 On Ambulatory Blood Pressure in Adults With Hypertension
Brief Title: Effect of PRM-125 on Ambulatory Blood Pressure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor
Sponsor: PRM Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-3001
Record Dates: First submitted 2022-01-02; First posted 2022-01-19 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRM125 (Experimental): PRM125
  Interventions: Drug: PRM-125

INTERVENTIONS:
Drug: PRM-125 — Antihypertensive

SUMMARY:
Evaluation of Once-Daily PRM125 On Ambulatory Blood Pressure in Adults with Hypertension

DETAILED DESCRIPTION:
Approximately 60 subjects with primary hypertension are treated for 8 weeks with PRM125 to determine if Ambulatory Blood Pressure is changed.

ELIGIBILITY:
Inclusion Criteria:

* primary hypertension

Exclusion Criteria:

* medical conditions that preclude evaluation and/or adversely effect subject safety

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour Systolic Blood Pressure | 8 weeks

SECONDARY OUTCOMES:
Change in 24 hour Diastolic Blood Pressure | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AMR, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No